CLINICAL TRIAL: NCT03350399
Title: The Relationship Between Second Trimester Placental Growth Factor Level and Fetal Growth Restriction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: amera mohamed (Other)
Responsible Party: Sponsor-Investigator, amera mohamed, professor, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: asamy
Record Dates: First submitted 2017-11-13; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Intra Uterine Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- level of placenta growth factor in IUGR
  Interventions: Diagnostic Test: placenta growth factor

INTERVENTIONS:
Diagnostic Test: placenta growth factor — estimation level of derum placenta growth factor

SUMMARY:
Type of the study:

A prospective observational study

Study settings:

The study will be conducted at Ain Shams University Maternity Hospital, Obstetrics and Gynecology Department, Faculty of medicine over a period of six month from July 2017 to December 2017.

Study population:

The study population comprises 60 pregnant women at 13 to 28 week of gestation attending outpatient clinic and emergency Ain Shams University Maternity Hospital, Obstetrics and Gynecology Department, Faculty of medicine.

Sample size justification Sample size was calculated using PASS 11.0 sample size calculation program and based on the study carried out by Benton, et al. (2016) Group sample sizes of 30 in group one (IUGR) and 30 in group two (Controls) achieve 80% power to detect a difference between the group proportions of 0.2910. The proportion in group one (the treatment group) is assumed to be 0.2940 under the null hypothesis and 0.5850 under the alternative hypothesis. The proportion in group two (the control group) is 0.2940. The test statistic used is the two-sided Z test with pooled variance. The significance level of the test was targeted at 0.0500. The significance level actually achieved by this design is 0.0506. The primary outcome is birth weight below the 10 the percentile. The sample size was inflated by 15.0% to account for lost to follow up (attrition problem).

Inclusion criteria:

Singleton pregnancy between 13-28 weeks of gestation. Pregnant women aged 18 - 35 years Pregnant women with fetal abdominal circumference (AC) < 10th percentile for gestational age (GA) on ultrasound

Exclusion criteria:

To exclude any factors that cause IUGR:

Chronic or gestational hypertension and/or preeclampsia Premature rupture of membranes A fetus with known chromosomal and/or congenital abnormalities confirmed after delivery.

Multiple gestation

DETAILED DESCRIPTION:
Full history: including age, gravidity, parity and gestational age Clinical examination: be physically examined. Abdominal examination and measurement of symphsis-fundal height Diagnosis of IUGR will be confirmed by ultrasound and confirmed by Doppler ultrasound of Umbilical artery and cerebral artery blood flow in 3rd trimester

ELIGIBILITY:
Inclusion Criteria:

- Singleton pregnancy between 13-28 weeks of gestation. Pregnant women aged 18 - 35 years Pregnant women with fetal abdominal circumference (AC) < 10th percentile for gestational age (GA) on ultrasound

Exclusion Criteria:

* Chronic or gestational hypertension and/or preeclampsia Premature rupture of membranes A fetus with known chromosomal and/or congenital abnormalities confirmed after delivery.

Multiple gestation

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population comprises 60 pregnant women at 13 to 28 week of gestation attending outpatient clinic and emergency Ain Shams University Maternity Hospital, Obstetrics and Gynecology Department, Faculty of medicine.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2017-12-20 (Estimated); Study Completion 2018-03-20 (Estimated)

PRIMARY OUTCOMES:
Birth weight below 10th percentile will be calculated as the primary outcome. | 2 month

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Sahms University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided